CLINICAL TRIAL: NCT02885987
Title: Use of Accessory Device AmplifEYE During Average Risk Screening Colonoscopy to Increase Adenoma Detection Rate
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: decided not to go ahead with study at this time
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Alexander Jahng, MD, Assistant Professor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 5160326
Record Dates: First submitted 2016-07-08; First posted 2016-09-01 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Standard Colonoscopy (No Intervention): AmplifEYE will not be used.
- Colonoscopy with AmplifEYE (Experimental): AmplifEYE accessory device will be attached to the colonoscope prior to starting the procedure
  Interventions: Device: AmplifEYE

INTERVENTIONS:
Device: AmplifEYE — AmplifEYE will be attached to the tip of the colonoscope prior to start of procedure.
  Other Names: colonoscope accessory device
  Arms: Colonoscopy with AmplifEYE

SUMMARY:
The purpose of this investigator-initiated study is to determine whether the use of an accessory device called AmplifEYE can improve colonoscopy quality in patients who are undergoing average risk colorectal cancer screening. Primary end point is adenoma detection rates.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients greater than or at 50 years of age who are referred for average risk screening colonoscopy.

Exclusion Criteria:

* Any pregnant patient
* Patient's that are unable to provide consent for themselves
* Any patient undergoing diagnostic colonoscopy (IBD, rectal bleeding, recent change in bowel habits, etc.)
* Any patient undergoing surveillance (prior history of polyps or colorectal cancer)
* Any patient undergoing high risk screening colonoscopy (family history of colon cancer in first degree family member <65 years of age, or co-existing conditions that pre-dispose to colon cancer such as polyposis syndromes, PSC or IBD)
* Prior history of any cancer
* Current or past immunosuppression (due to either infection or medications)
* Coagulation disorder OR use of anti-coagulation or anti-platelet therapy other than aspirin within 5-7 days of procedure
* Colonic strictures
* suspected intestinal obstruction or colonic pseudo-obstruction
* history of colon resection
* active infection
* active inflammation (including diverticulitis)

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-03 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Difference in adenoma detection rate (ADR), with and without use of AmplifEYE. | 1 week
  ADR is calculated by dividing the total number of screening procedures in which 1 or more histologically confirmed adenomas were detected by the total number of screening procedures performed.

SECONDARY OUTCOMES:
ADR will be differentiated according to morphology | 1 week
  ADR will be differentiated according to morphology (flat, sessile, pedunculated)
ADR will be differentiated according to final pathology | 1 week
  ADR will be differentiated according to final pathology (sessile serrated adenomas, traditional serrated polyps, tubular/villous adenomas)
ADR will be differentiated according to location | 1 week
  Location will be specified by colon segment and flexures.
Advanced ADR | 1 week
  calculated as same for ADR, but only in those with polyps that are >=1 cm in size, with components of villous features, or with those of dysplasia
Mean total number of polyps detected | 1 week
  calculated by dividing the total number of adenomas detected by the total number of screening procedures performed
ADR-plus | 1 week
  mean number of adenomas found after the first in procedures in which 1 or more adenomas were detected
APP (adenomas per positive participant) | 1 week
  calculated as the total number of adenomas detected during the first colonoscopy divided by the number of positive participants (those with ≥1 adenoma detected during the first colonoscopy)
APC (adenomas per colonoscopy) | 1 week
  calculated as the total number of adenomas detected during the first colonoscopy divided by the number of first colonoscopies
Quality metrics: time of colonoscopy | 1 hour
  Differences in quality metrics will be noted: cecal intubation time and total withdrawal time.
Quality metrics: prep quality | 1 hour
  Differences in prep quality will be noted
Sedative Medications used | 1 hour
  Differences in sedative medications used

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Jahng, MD, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No